CLINICAL TRIAL: NCT00000986
Title: A Safety, Tolerance, and Immunological Study of a Combination of Recombinant Interleukin 2 and Zidovudine in Patients With AIDS or AIDS Related Complex
Brief Title: The Safety and Effectiveness of Interleukin-2 Plus Zidovudine in Patients With AIDS or AIDS Related Complex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 067; 11041 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; Interleukin-2; Drug Interactions; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; aldesleukin

INTERVENTIONS:
Drug: Zidovudine
Drug: Aldesleukin

SUMMARY:
To test the safety and tolerance of three different doses of recombinant human interleukin 2 (aldesleukin; IL-2), when it is given for five consecutive days to patients with AIDS or AIDS related complex (ARC), who have also received zidovudine (AZT) for at least 6 weeks just before beginning the IL-2 treatment.

AZT is an antiviral drug, which has been shown to be beneficial in some patients with AIDS. IL-2 is a substance found naturally in the body that boosts the body's immune response to invading organisms and tumor cells. These two drugs, when administered together, may have a mutually helpful effect in treating AIDS patients, but before this effect can be studied, it is important to understand the proper dose and any side effects that may occur when these drugs are used together. The study will show how much AZT and IL-2 patients can safely take at the same time and how the two drugs will interact with each other.

DETAILED DESCRIPTION:
AZT is an antiviral drug, which has been shown to be beneficial in some patients with AIDS. IL-2 is a substance found naturally in the body that boosts the body's immune response to invading organisms and tumor cells. These two drugs, when administered together, may have a mutually helpful effect in treating AIDS patients, but before this effect can be studied, it is important to understand the proper dose and any side effects that may occur when these drugs are used together. The study will show how much AZT and IL-2 patients can safely take at the same time and how the two drugs will interact with each other.

AMENDED: Note that the dose of AZT changed 900214 to reflect new dose recommendations. Original design: Six weeks before beginning treatment with IL-2, patients are given AZT daily. There are three patient groups, one for each dose level of IL-2. On the first day of treatment with the two drugs together, patients are admitted to Presbyterian University Hospital, where AZT is administered orally every 4 hours and IL-2 is given once a day as a single injection under the skin. Clinical and laboratory safety data from the first two patients enrolled in each treatment group will be analyzed prior to enrolling additional patients in each group. All patients are expected to stay in the hospital for at least 5 days, and some may stay longer if serious side effects develop. AZT treatment will continue after the patient leaves the hospital for an additional 10 weeks. Follow-up visits are scheduled for days 6, 8, and 15 for safety, immunologic, and virologic evaluations. Thereafter, patients are followed by telephone interview every other week and come into the clinic if a change in health is reported. At weeks 10 and 20, patients are also evaluated in a follow-up clinic visit.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Acetaminophen under the supervision of a study physician.

Prior Medication:

Required for at least 6 weeks prior to study entry:

* Zidovudine at a dose of at least 300 mg/day.
* Allowed:
* Aerosolized pentamidine prior to combination therapy.

Patients must demonstrate the following clinical and laboratory findings:

* Currently receiving zidovudine (AZT) at a dose of at least 300 mg/day and have received the drug for at least 6 weeks.
* Have a life expectancy of = or > 4 months.
* Available for the duration of the study and for follow-up visits.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions will be excluded:

* Evidence of active life-threatening opportunistic infection with bacterial, viral, fungal, or protozoan pathogens during the 6-week period prior to and during the 5-day period of combination therapy.
* A fever > 101 degrees F within the past 10 days.
* Significant central nervous system disease, including acquired immunodeficiency syndrome (AIDS), dementia, psychiatric disabilities, or seizure disorders.
* Significant cardiac (New York Heart Association stage III or IV) and/or pulmonary disease (forced expiratory volume < 75 percent).
* Kaposi's sarcoma or other AIDS related malignancy.
* Evidence of malabsorption as indicated by 10 percent weight loss within the last 3 months.

Concurrent Medication:

Excluded:

* Cardiac medications.
* Glucocorticosteroids.
* Probenecid.
* Acetylsalicylic acid.
* Trimethoprim / sulfamethoxazole.
* Acyclovir.
* Allopurinol.
* Drugs causing anemia, neutropenia, or nephrotoxicity.
* Aerosolized pentamidine during combination therapy.
* Nonsteroidal anti-inflammatory drugs by patients with thrombocytopenia (<75000 platelets/mm3).
* Acetaminophen except under supervision of a study physician.

Patients with the following conditions will be excluded:

* Evidence of active life-threatening opportunistic infection with bacterial, viral, fungal, or protozoan pathogens during the 6-week period prior to and during the 5-day period of combination therapy.
* A fever > 101 degrees F within the past 10 days.
* Significant central nervous system disease, including acquired immunodeficiency syndrome (AIDS), dementia, psychiatric disabilities, or seizure disorders.
* Significant cardiac (New York Heart Association stage III or IV) and/or pulmonary disease (forced expiratory volume < 75 percent).
* Kaposi's sarcoma or other AIDS related malignancy.
* Evidence of malabsorption as indicated by 10 percent weight loss within the last 3 months.

Prior Medication:

Excluded within 4 weeks of study entry:

* Any antiretroviral drug, except zidovudine (AZT).
* Excluded within 12 weeks of study entry:
* Immunotherapy, including interleukins, interferons, tumor necrosis factor.
* Other cytokines.
* Biologic response modifiers.
* Monoclonal antibodies.
* BCG vaccines.

Active drug or alcohol abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18
Dates: Study Completion 1994-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Ho, Study Chair
Locations (1):
- Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] McMahon DK, Armstrong JA, Huang XL, Rinaldo CR Jr, Gupta P, Whiteside TL, Pazin GJ, Tripoli C, Ho M. A phase I study of subcutaneous recombinant interleukin-2 in patients with advanced HIV disease while on zidovudine. AIDS. 1994 Jan;8(1):59-66. doi: 10.1097/00002030-199401000-00009. PMID 8011237